CLINICAL TRIAL: NCT02758613
Title: A Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3009104 in Healthy Chinese Subjects
Brief Title: A Study of Baricitinib (LY3009104) in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14778; I4V-GH-JAGR (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-04-29; First posted 2016-05-02 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-07

CONDITIONS: Healthy
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 milligram (mg) Baricitinib (Experimental): 2mg Baricitinib administered orally, once on Day 1 and once a day (QD) on Days 4 through 10 (7 days).
  Interventions: Drug: Baricitinib
- 4mg Baricitinib (Experimental): 4mg Baricitinib administered orally, once on Day 1 and QD on Days 4 through 10 (7 days).
  Interventions: Drug: Baricitinib
- 10mg Baricitinib (Experimental): 10mg Baricitinib administered orally, once on Day 1 and QD on Days 4 through 10 (7 days).
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Placebo matching Baricitinib administered orally, once on Day 1 and QD on Days 4 through 10 (7 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: 10mg Baricitinib; 2 milligram (mg) Baricitinib; 4mg Baricitinib
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the safety and tolerability of the study drug known as baricitinib in healthy Chinese participants. The study will measure how the body absorbs, breaks down and gets rid of baricitinib. The study will last about 20 days, not including screening. This study is for research purposes only, and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy Chinese males agreed to use methods of birth control or are postmenopausal Chinese females, as determined by medical history and physical examination
* Have a body mass index of 19.0 to 24.0 kilograms per meter squared (kg/m²), inclusive, at screening.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.

Exclusion Criteria:

* Have a history of adverse drug reactions or "drug allergy" to more than 3 types of systemically administered medications.
* Have an abnormality in the 12-lead electrocardiogram (ECG).
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history of stomach or intestinal surgery.
* Current or recent history (<30 days prior to screening of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection.
* Have an absolute neutrophil count (ANC) less than 2000 cell/microliter (μL) (2 x 109/liter [L]).
* Have current herpes zoster or simplex within 90 days prior to the first dose,
* Have evidence of active or latent tuberculosis (TB)
* Have used or intend to use over-the-counter, prescription medication, or Chinese herbal preparation within 14 days prior to dosing and during the study.
* Have consumed grapefruit, grapefruit juice, or grapefruit products within 7 days prior to the first dose or are unwilling to abide by the grapefruit restrictions during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- 2mg Baricitinib: 2mg baricitinib administered orally, once on Day 1 and QD on Days 4 through 10 (7 days).
Period: Treatment
Arm/Group | Placebo | 2mg Baricitinib | 4mg Baricitinib | 10mg Baricitinib
Started | 8 | 8 | 9 | 8
Received at Least One Dose of Study Drug | 8 | 8 | 9 | 8
Completed | 6 | 8 | 8 | 8
Not Completed | 2 | 0 | 1 | 0
Not completed — Physician and Sponsor Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Period: Follow-up
Arm/Group | Placebo | 2mg Baricitinib | 4mg Baricitinib | 10mg Baricitinib
Started | 6 | 8 | 8 | 8
Completed | 6 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Placebo matching baricitinib administered orally, once on Day 1 and once a day (QD) on Days 4 through 10 (7 days).
- 2mg Baricitinib: 2mg baricitinib administered orally, once on Day 1 and once a day (QD) on Days 4 through 10 (7 days).
- 4mg Baricitinib: 4mg baricitinib administered orally, once on Day 1 and once a day (QD) on Days 4 through 10 (7 days).
- 10mg Baricitinib: 10mg baricitinib administered orally, once on Day 1 and once a day (QD) on Days 4 through 10 (7 days).
- Total: Total of all reporting groups
Arm/Group | Placebo | 2mg Baricitinib | 4mg Baricitinib | 10mg Baricitinib | Total
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (5.4) | 30.8 (7.3) | 26.6 (3.5) | 27.6 (6.7) | 27.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 9 | 8 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 9 | 8 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 8 | 8 | 9 | 8 | 33
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 22.34 (1.21) | 22.15 (1.75) | 21.87 (1.28) | 21.68 (1.39) | 22.01 (1.38)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Clinically Significant Event(s)
Description: Clinically significant events were defined as a moderate to severe adverse event, abnormal clinical sign, or clinical laboratory finding that may pose risk to the well-being of the participant. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through Study Completion (up to Day 20)
Population: All randomized participants who received at least one dose of study drug and experienced clinically significant event.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 2mg Baricitinib | 4mg Baricitinib | 10mg Baricitinib
Number analyzed (Participants) | 8 | 8 | 9 | 8
Participants | 4 | 0 | 2 | 4

2. Secondary Outcome: Pharmacokinetics(PK): Maximum Concentration (Cmax) of Baricitinib
Description: Maximum observed drug concentration for single dose and Cmax as steady date for multiple dosing.
Time Frame: Day 1: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Postdose; Day 5: Predose; Day 6: Predose; Day 7: Predose; Day 8: Predose; Day 9: Predose; Day 10: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Postdose
Population: All randomized participants who received at least one dose of baricitinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 2mg Baricitinib | 4mg Baricitinib | 10mg Baricitinib
Number analyzed (Participants) | 8 | 9 | 8
nanogram per milliliter (ng/mL)
  Single Dose Day 1 | 24.3 (17) | 47.8 (42) | 147 (28)
  Multiple Dose Day 10: number analyzed (Participants) | 8 | 8 | 8
  Multiple Dose Day 10 | 28.0 (24) | 48.0 (28) | 136 (17)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of Baricitinib
Description: Area under the concentration versus time curve from zero to infinity (AUC0-inf) during single dose and area under the concentration versus time curve (AUCtau,ss) during multiple dose of baricitinib at steady state.
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of baricitinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram * hour per milliliter (ng*h/mL)
Arm/Group | 2mg Baricitinib | 4mg Baricitinib | 10mg Baricitinib
Number analyzed (Participants) | 8 | 9 | 8
nanogram * hour per milliliter (ng*h/mL)
  Single Dose Day 1: number analyzed (Participants) | 8 | 8 | 8
  Single Dose Day 1 | 139 (12) | 270 (17) | 777 (9)
  Multiple Dose Day 10: number analyzed (Participants) | 8 | 8 | 8
  Multiple Dose Day 10 | 145 (12) | 265 (18) | 771 (14)

ADVERSE EVENTS:
Arm/Group | Placebo | 2mg Baricitinib | 4mg Baricitinib | 10mg Baricitinib
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 1/8 | 2/9 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 2mg Baricitinib (N=8) | 4mg Baricitinib (N=9) | 10mg Baricitinib (N=8)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days